CLINICAL TRIAL: NCT02942160
Title: A Phase 2, Open-Label Extension Study of EN3835 in the Treatment of Edematous Fibrosclerotic Panniculopathy
Brief Title: EN3835 for the Treatment of Edematous Fibrosclerotic Panniculopathy (Commonly Known as Cellulite)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3835-202
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Edematous Fibrosclerotic Panniculopathy; Cellulite
MeSH Terms: conditions — Cellulite | interventions — Microbial Collagenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EN3835 Active (Experimental): EN3835 0.84mg (Collagenase Clostridium Histolyticum)
  Interventions: Biological: Collagenase Clostridium Histolyticum

INTERVENTIONS:
Biological: Collagenase Clostridium Histolyticum
  Other Names: Xiaflex

SUMMARY:
A Phase 2, Open-Label Extension Study of EN3835 in the Treatment of Edematous Fibrosclerotic Panniculopathy (commonly known as Cellulite).

ELIGIBILITY:
Inclusion Criteria for Observation Phase:

* Voluntarily sign and date an informed consent agreement
* Have participated in and completed the double-blind study EN3835-201
* Be willing to apply sunscreen to any treated quadrant before each exposure to sun

Inclusion Criteria for Treatment Phase:

* Voluntarily sign and date an informed consent agreement
* Have participated in and completed the double-blind study EN3835-201
* Be willing to apply sunscreen to any treated quadrant before each exposure to sun
* Have at least 1 quadrant with: a score of 3 or 4 (moderate or severe) as reported on the PCSS (Photonumeric Cellulite Severity Scale) by the subject or investigator, and a Hexsel CSS (Cellulite Severity Scale) score no greater than 13
* Be judged to be in good health
* Have a negative urine pregnancy test at screening and be using an effective contraception method, be surgically sterile, or post-menopausal

Exclusion Criteria for Observation Phase:

* None

Exclusion Criteria for Treatment Phase:

* Has used, or intends to use during the course of the study, other treatment of EFP on the legs or buttocks
* Is presently nursing a baby or providing breast milk for a baby
* Intends to become pregnant during the study
* Currently receiving, has received within 7 days before injection of study drug, or plans to receive an anticoagulant or antiplatelet medication
* History of stroke or bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mike McLane, Study Director — Endo Pharmaceuticals
Locations (15):
- United States (15):
  - Endo Clinical Trial Site #1, Beverly Hills, California
  - Endo Clinical Trial Site #2, Murrieta, California
  - Endo Clinical Trial Site #3, Oceanside, California
  - Endo Clinical Trial Site #4, San Diego, California
  - Endo Clinical Trial Site #5, Clearwater, Florida
  - Endo Clinical Trial Site #6, Coral Gables, Florida
  - Endo Clinical Trial Site #7, Palm Beach, Florida
  - Endo Clinical Trial Site #8, Washington, Missouri
  - Endo Clinical Trial Site #10, New York, New York
  - Endo Clinical Trial Site #9, New York, New York
  - Endo Clinical Trial Site #11, Nashville, Tennessee
  - Endo Clinical Trial Site #12, Pflugerville, Texas
  - Endo Clinical Trial Site #13, Charlottesville, Virginia
  - Endo Clinical Trial Site #14, Lynchburg, Virginia
  - Endo Clinical Trial Site #15, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- EN3835 Treated Participants in EN3835-202: Observation Phase (259 Started & 222 Completed):
  Observation of Buttock or Thigh Treated with EN3835: 0.84mg Collagenase Clostridium Histolyticum or with Placebo in Study EN3835-201
  EN3835 Treated Participants in EN3835-202:
  Buttock & Thigh Treatment Regions Treated with EN3835 0.84mg Collagenase Clostridium Histolyticum
Period: Overall Study
Arm/Group | EN3835 Treated Participants in EN3835-202
Started | 259 (Observation Phase prior to open-label treatment phase)
EN3835-202 Participants | 222 (Observation Phase Completed)
EN3835 Treated Subjects in EN3835-202 | 200 (EN3835 Treated Participants in EN3835-202 Started)
Completed | 156 (EN3835 Treated Participants in EN3835-202 Completed)
Not Completed | 103

BASELINE CHARACTERISTICS:
Groups:
- EN3835 Treatment Regions: Buttock & Thigh Treatment Regions Treated with EN3835 0.84mg Collagenase Clostridium Histolyticum
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (11.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46
  Not Hispanic or Latino | 154
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 25
  White | 173
  More than one race | 0
  Unknown or Not Reported | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.3 (6.78)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Were 2-level Composite (CR-PCSS and PR-PCSS) Responders During the Observation Phase
Description: Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) and Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS) is a 5-level scale ranging from "0" (None) to "4" (Severe). A 2-level composite responder is a participant that received EN3835 with a reduction (decrease in score) in severity of at least 2-levels from baseline on both the CR-PCSS and the PR-PCSS at a particular visit.
  Observation Phase is defined as the time period from Screening to the first treatment date of the same treatment area in Study EN3835-202, or the end of Study EN3835-202 if there was no treatment received for the same treatment area in Study EN3835-202. Three participants were discontinued from the study after Day 180, percentages are based on the observed counts.
Time Frame: Day 180 to Day 360
Population: The Durability Population for Double-blind Treated Participants is defined as all participants in the Overall Durability Population for both who showed an improvement on Day 71 of at least 2-level on each scale (CR-PCSS and PR-PCSS) from the baseline for the treatment area treated with EN3835 in the double-blind study (EN3835-201).
Measure: Count of Participants; unit: Participants
Groups:
- EN3835 Treatment Regions: Buttocks & Thighs Treated with EN3835: 0.84mg Collagenase Clostridium Histolyticum
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 19
Participants
  Observation Visit Day 180: Yes | 19
  Observation Visit Day 180: No | 0
  Observation Visit Day 360: number analyzed (Participants) | 16
  Observation Visit Day 360: Yes | 16
  Observation Visit Day 360: No | 0

2. Secondary Outcome: Number of Participants That Were 1-level Composite (CR-PCSS and PR-PCSS) Responders During the Observation Phase
Description: Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) and Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS) is a 5-level scale ranging from "0" (None) to "4" (Severe). A 1-level composite responder is a participant that received EN3835 with a reduction (decrease in score) in severity of at least 1-level from baseline on both the PR-PCSS and the CR-PCSS at a particular visit. Observation Phase is defined as the time period from Screening to the first treatment date of the same treatment area in Study EN3835-202, or the end of Study EN3835-202 if there was no treatment received for the same treatment area in Study EN3835-202.
Time Frame: Day 180 to Day 360
Population: The Durability Population for Double-blind Treated Participants is defined as all participants in the Overall Durability Population who showed an improvement on Day 71 of at least 1-level on each scale (CR-PCSS and PR-PCSS) from the baseline for the treatment area treated with EN3835 in the double-blind study (EN3835-201).
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 53
Participants
  Observation Durability Visit Day 180: Yes | 50
  Observation Durability Visit Day 180: No | 3
  Observation Durability Visit Day 360: number analyzed (Participants) | 45
  Observation Durability Visit Day 360: Yes | 43
  Observation Durability Visit Day 360: No | 2

3. Secondary Outcome: Number of Participants That Were 2-level Composite (CR-PCSS and PR-PCSS) Responders During the Long-term Durability Phase
Description: Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) and Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS) is a 5-level scale ranging from "0" (None) to "4" (Severe). A 2-level composite responder is a participant that received EN3835 with a reduction (decrease in score) in severity of at least 2-levels from baseline on both the CR-PCSS and the PR-PCSS at a particular visit. Long-term Durability Phase is defined as all participants in the Overall Durability Population who showed an improvement on Day 71 of at least 1-level on each scale (CR-PCSS and PR-PCSS) from baseline for the treatment area treated with EN3835 in the double-blind Study (EN3835-201).
Time Frame: Day 540 to Day 720
Population: The Durability Population for Double-blind Treated Participants, defined as all participants who showed an improvement on Day 71 of at least 2-level on each scale (CR-PCSS and PR-PCSS) from the baseline for the treatment area treated with EN3835 in the double-blind study (EN3835-201), and had an Observation at Day 540.
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 7
Participants
  Long-term Durability Visit Day 540: Yes | 7
  Long-term Durability Visit Day 540: No | 0
  Long-term Durability Visit Day 720: Yes | 7
  Long-term Durability Visit Day 720: No | 0

4. Secondary Outcome: Number of Participants That Were 1-level Composite (CR-PCSS and PR-PCSS) Responders During the Long-term Durability Phase
Description: Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) and Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS) is a 5-level scale ranging from "0" (None) to "4" (Severe). A 1-level composite responder is a participant who received EN3835 with a reduction (decrease in score) in severity of at least 1-level from baseline on both the PR-PCSS and the CR-PCSS at a particular visit. Long-term Durability Phase is defined as all participants in the Overall Durability Population who showed an improvement on Day 71 of at least 1-level on each scale (CR-PCSS and PR-PCSS) from baseline for the treatment area treated with EN3835 in the double-blind Study (EN3835-201).
Time Frame: Day 540 to Day 720
Population: The Durability Population for Double-blind Treated Participants, defined as all participants who showed an improvement on Day 71 of at least 1-level on each scale (CR-PCSS and PR-PCSS) from the baseline for the treatment area treated with EN3835 in the double-blind study (EN3835-201), and had an Observation at Day 540.
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 23
Participants
  Long-term Durability Visit Day 540: Yes | 22
  Long-term Durability Visit Day 540: No | 1
  Long-term Durability Visit Day 720: Yes | 21
  Long-term Durability Visit Day 720: No | 2

5. Secondary Outcome: CR-PCSS Change From Baseline (in EN3835-201 Study) by Visit During the Observation Phase
Description: Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) is a 5-level scale ranging from "0" (None) to "4" (Severe). A negative change from baseline indicates an improvement in cellulite severity. Observation Phase is defined as the time period from Screening to the first treatment date of the same treatment area in Study EN3835-202, or the end of Study EN3835-202 if there was no treatment received for the same treatment area in Study EN3835-202.
Time Frame: Baseline (in EN3835-201 Study) to Observation Day 360
Population: Observation Population included all participants who rolled over from Study EN3835-201 (all 259 participants that rolled over in Observation Phase).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- EN3835 0.84 mg: Treatment in Study EN3835-201
- Placebo: Placebo in Study EN3835-201
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 121 | 138
score on a scale
  Change from Baseline on Day 71 (EN3835-201 Study) | -0.8 (0.88) | -0.3 (0.60)
  Change from Baseline-Observation Visit Day 180: number analyzed (Participants) | 120 | 137
  Change from Baseline-Observation Visit Day 180 | -0.6 (0.80) | -0.2 (0.67)
  Change from Baseline-Observation Visit Day 270: number analyzed (Participants) | 106 | 89
  Change from Baseline-Observation Visit Day 270 | -0.6 (0.76) | -0.1 (0.63)
  Change from Baseline-Observation Visit Day 360: number analyzed (Participants) | 97 | 20
  Change from Baseline-Observation Visit Day 360 | -0.9 (0.86) | -0.5 (0.83)

6. Secondary Outcome: CR-PCSS Change From Baseline (BL) by Visit During the Treatment Phase for Participants With a Second EN3835 Treatment
Description: Clinician-Reported Photonumeric Cellulite Severity Scale (CR-PCSS) is a 5-level scale ranging from "0" (None) to "4" (Severe). A decrease in the CR-PCSS score from baseline indicates an improvement in cellulite severity. Treatment phase is defined as the time period from the second EN3835 treatment date to the end of Study EN3835-202. One hundred sixty-two participants received a second treatment course Study EN3835-202 and were included in the Effectiveness Population. This retreated/redosed treatment group comprised 87 participants that received their second treatment course of EN3835 in Study EN3835-202 having received their first treatment course in Study EN3835-201 and 75 participants that received both their first and second treatment courses in Study EN3835-202.
Time Frame: Day 22 to Day 360
Population: Effectiveness Population included all safety participants who had a baseline and at least 1 post-baseline assessment on both the CR-PCSS and PR-PCSS on the treatment area selected for treatment in Study EN3835-202.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 162
score on a scale
  Change from Baseline (BL) to Treatment Day 22: number analyzed (Participants) | 154
  Change from Baseline (BL) to Treatment Day 22 | -0.6 (0.68)
  Change from Baseline (BL) to Treatment Day 43: number analyzed (Participants) | 160
  Change from Baseline (BL) to Treatment Day 43 | -0.8 (0.71)
  Change from Baseline (BL) to Treatment Day 71: number analyzed (Participants) | 159
  Change from Baseline (BL) to Treatment Day 71 | -1.0 (0.79)
  Change from BL to Treatment Observation Day 180: number analyzed (Participants) | 154
  Change from BL to Treatment Observation Day 180 | -1.0 (0.80)
  Change from BL to Treatment Observation Day 360: number analyzed (Participants) | 142
  Change from BL to Treatment Observation Day 360 | -0.9 (0.77)

7. Secondary Outcome: PR-PCSS Change From Baseline by Visit in Treatment Phase for Participants With Second EN3835 Treatment
Description: Patient-Reported Photonumeric Cellulite Severity Scale (PR-PCSS) is a 5-level scale ranging from "0" (None) to "4" (Severe). A decrease in the PR-PCSS score from baseline indicates an improvement in cellulite severity. Treatment phase is defined as the time period from the second EN3835 treatment date to the end of Study EN3835-202. One hundred sixty-two participants received a second treatment course in this study and were included in the Effectiveness Population. This retreated/redosed treatment group comprised 87 participants that received their second treatment course of EN3835 in Study EN3835-202 having received their first treatment course in Study EN3835-201 and 75 participants that received both their first and second treatment courses in Study EN3835-202.
Time Frame: Day 22 to Day 360
Population: Effectiveness Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 162
score on a scale
  Change from Baseline (BL) to Treatment Day 22: number analyzed (Participants) | 154
  Change from Baseline (BL) to Treatment Day 22 | -0.5 (0.64)
  Change from Baseline (BL) to Treatment Day 43: number analyzed (Participants) | 160
  Change from Baseline (BL) to Treatment Day 43 | -0.8 (0.75)
  Change from Baseline (BL) to Treatment Day 71: number analyzed (Participants) | 159
  Change from Baseline (BL) to Treatment Day 71 | -1.1 (0.82)
  Change from BL to Treatment Observation Day 180: number analyzed (Participants) | 155
  Change from BL to Treatment Observation Day 180 | -1.0 (0.83)
  Change from BL to Treatment Observation Day 360: number analyzed (Participants) | 143
  Change from BL to Treatment Observation Day 360 | -1.0 (0.83)

8. Secondary Outcome: Change From Baseline on the Hexsel CSS Total Score During the Observation Phase
Description: The Hexsel Cellulite Severity Scale (CSS) is a photonumeric scale that evaluates 5 key morphologic features of cellulite: (A) number of evident depressions, (B) depth of depressions, (C) morphological appearance of skin surface alterations, (D) laxity, flaccidity or sagging of skin, and (E) current classification scale based on medical literature. Each of these features is evaluated on a 4-point scale from a low of "0" to a high of "3", with higher scores signifying more severe cellulite. The Hexcel CSS total score is the sum of all 5 features and can range from "0" (no cellulite) to "15" (extremely severe cellulite) and is designated in this study as the Hexsel CSS total score.
Time Frame: Baseline (in EN3835-201 Study) to Day 360
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 121 | 138
score on a scale
  Baseline Point (in EN3835-201 Study) | 10.7 (1.32) | 10.4 (1.41)
  Day 71 Reference Point (in EN3835 Study) | 9.0 (2.42) | 9.7 (2.20)
  Change from Baseline (Day 71) | -1.8 (2.22) | -0.8 (1.81)
  Observation Visit Day 360: number analyzed (Participants) | 97 | 19
  Observation Visit Day 360 | 8.6 (2.40) | 9.5 (1.35)
  Change from Baseline (Day 360): number analyzed (Participants) | 97 | 19
  Change from Baseline (Day 360) | -2.2 (2.34) | -1.2 (1.47)

9. Secondary Outcome: Change From Baseline (BL) in the Hexsel CSS Total Score During Long-term Durability Visits
Description: The Hexsel Cellulite Severity Scale (CSS) is a photonumeric scale that evaluates 5 key morphologic features of cellulite: (A) number of evident depressions, (B) depth of depressions, (C) morphological appearance of skin surface alterations, (D) laxity, flaccidity or sagging of skin, and (E) current classification scale based on medical literature. Each of these features is evaluated on a 4-point scale from a low of "0" to a high of "3", with higher scores indicating more severe cellulite. The total score is a summation of all 5 features and can range from "0" (no cellulite) to "15" (extremely severe cellulite) and is designated in this study as the Hexsel CSS total score. A negative change from baseline indicates an improvement in cellulite severity.
Time Frame: Day 540 to Day 720
Population: Durability Population in Double-blind Treated Participants is defined as all participants in the Overall Durability Population who showed an improvement on Day 71 of at least 1-level on each scale (CR-PCSS and PR-PCSS) from the baseline for the treatment area treated with EN3835 in the double-blind study (EN3835-201).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 53
score on a scale
  Baseline (in EN3835-201 Study) | 10.6 (1.43)
  Long-term Durability Visit Day 540-Change from BL: number analyzed (Participants) | 6
  Long-term Durability Visit Day 540-Change from BL | -3.5 (1.76)
  Long-term Durability Visit Day 720-Change from BL: number analyzed (Participants) | 23
  Long-term Durability Visit Day 720-Change from BL | -2.9 (1.74)

10. Secondary Outcome: Change From Baseline in Hexsel CSS Total Score in Treatment Phase for Participants With Second EN3835 Treatment
Description: The Hexsel Cellulite Severity Scale (CSS) is a photonumeric scale that evaluates 5 key morphologic features of cellulite: (A) number of evident depressions, (B) depth of depressions, (C) morphological appearance of skin surface alterations, (D) laxity, flaccidity or sagging of skin, and (E) current classification scale based on medical literature. Each of these features is evaluated on a 4-point scale from a low of "0" to a high of "3". The total score is a summation of all 5 features and can range from "0" (no cellulite) to "15" (extremely severe cellulite) and is designated in this study as the Hexsel CSS total score. Change from baseline is the visit total score minus baseline total score. A negative change from baseline indicates an improvement in cellulite severity.
  Treatment phase is defined as the time period from the second EN3835 treatment date to the end of Study EN3835-202.
Time Frame: Baseline - Day 360
Population: Effectiveness Population included all safety participants who had a baseline and at least 1 post-baseline assessment on both the CR-PCSS and PR-PCSS on the treatment area selected for treatment in the current study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 162
score on a scale
  Second EN3835 Treatment: Baseline | 10.5 (1.44)
  Second EN3835 Treatment: Day 71: number analyzed (Participants) | 159
  Second EN3835 Treatment: Day 71 | 8.3 (2.41)
  Second EN3835 Treatment: Change from Baseline: number analyzed (Participants) | 159
  Second EN3835 Treatment: Change from Baseline | -2.2 (2.32)
  Second EN3835: Treatment Observation Day 360: number analyzed (Participants) | 143
  Second EN3835: Treatment Observation Day 360 | 8.1 (2.51)
  Second EN3835: Change from Baseline: number analyzed (Participants) | 143
  Second EN3835: Change from Baseline | -2.4 (2.37)

11. Secondary Outcome: Investigator Global Aesthetic Improvement Scale (I-GAIS) at Observation Visit Day 360 During the Observation Phase
Description: Investigator Global Aesthetic Improvement Scale (I-GAIS) is a 7-point numeric scale that evaluates the improvement of the treated treatment area in global aesthetics. The scale ranges from "+3" (Very much improved) to "-3" (Very much worse), an increase in the I-GAIS scores indicates an improvement in Global Aesthetic Score. Percentages are based on the number of all evaluable subjects at each visit. Observation Phase is defined as the time period from Screening to the first treatment date of the same treatment area in Study EN3835-202, or the end of Study EN3835-202 if there was no treatment received for the same treatment area in Study EN3835-202.
Time Frame: Day 360
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 97 | 19
Participants
  Very Much Improved (3) | 4 | 0
  Much Improved (2) | 23 | 0
  Improved (1) | 36 | 4
  No Change (0) | 32 | 14
  Worse (-1) | 2 | 1
  Much Worse (-2) | 0 | 0
  Very Much Worse (-3) | 0 | 0

12. Secondary Outcome: Investigator Global Aesthetic Improvement Scale (I-GAIS) in Treatment Phase for Participants With Second EN3835 Treatment
Description: Investigator Global Aesthetic Improvement Scale (I-GAIS) is a 7-point numeric scale that evaluates the improvement of the treated treatment area in global aesthetics. The scale ranges from "+3" (Very much improved) to "-3" (Very much worse), an increase in the I-GAIS indicates an improvement in global aesthetics. Percentages are based on the number of all evaluable participants at each visit. One hundred sixty-two participants received a second treatment course in this study and were included in the Effectiveness Population. This retreated/dosed treatment group comprised 87 participants that received their second treatment course of EN3835 in Study EN3835-202 having received their first treatment course in Study EN3835-201 and 75 participants that received both their first and second treatment course in Study EN3835-202.
Time Frame: Day 71 - Day 360
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 162
Participants
  Second EN3835 Treatment: Treatment Day 71: number analyzed (Participants) | 159
  Second EN3835 Treatment: Treatment Day 71: Very Much Improved (3) | 10
  Second EN3835 Treatment: Treatment Day 71: Much Improved (2) | 38
  Second EN3835 Treatment: Treatment Day 71: Improved (1) | 73
  Second EN3835 Treatment: Treatment Day 71: No Change (0) | 35
  Second EN3835 Treatment: Treatment Day 71: Worse (-1) | 3
  Second EN3835 Treatment: Treatment Day 71: Much Worse (-2) | 0
  Second EN3835 Treatment: Treatment Day 71: Very Much Worse (-3) | 0
  Second EN3835 Tx: Treatment Observation Day 360: number analyzed (Participants) | 142
  Second EN3835 Tx: Treatment Observation Day 360: Very Much Improved (3) | 5
  Second EN3835 Tx: Treatment Observation Day 360: Much Improved (2) | 33
  Second EN3835 Tx: Treatment Observation Day 360: Improved (1) | 64
  Second EN3835 Tx: Treatment Observation Day 360: No Change (0) | 31
  Second EN3835 Tx: Treatment Observation Day 360: Worse (-1) | 7
  Second EN3835 Tx: Treatment Observation Day 360: Much Worse (-2) | 2
  Second EN3835 Tx: Treatment Observation Day 360: Very Much Worse (-3) | 0

13. Secondary Outcome: Subject Global Aesthetic Improvement Scale (S-GAIS) at the End of Study (EOS) During the Observation Phase, Observation Visit Day 360
Description: Subject Global Aesthetic Improvement Scale (S-GAIS) is a 7-point numeric scale that evaluates the improvement of the treated treatment area in global aesthetics. The scale ranges from "+3" (Very much improved) to "-3" (Very much worse), an increase in S-GAIS indicates an improvement. Percentages are based on the number of all evaluable participants at each visit. Observation Phase is defined as the time period from Screening to the first treatment date of the same treatment area in Study EN3835-202, or the end of Study EN3835-202 if there was no treatment received for the same treatment area in Study EN3835-202.
Time Frame: Day 360
Population: Observation Population included all participants who rolled over from Study EN3835-201
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 97 | 19
Participants
  Very Much Improved (3) | 3 | 0
  Much Improved (2) | 18 | 0
  Improved (1) | 46 | 4
  No Change (0) | 23 | 14
  Worse (-1) | 5 | 1
  Much Worse (-2) | 0 | 0
  Very Much Worse (-3) | 2 | 0

14. Secondary Outcome: Subject Global Aesthetic Improvement Scale (S-GAIS) During the Treatment Phase for Participants With Second EN3835 Treatment
Description: Subject Global Aesthetic Improvement Scale (S-GAIS) is a 7-point numeric scale that evaluates the improvement of the treated treatment area in global aesthetics. The scale ranges from "+3" (Very much improved) to "-3" (Very much worse). Percentages are based on the number of evaluable participants at each visit. One hundred sixty-two participants received a second treatment course in EN3835-202 Study and were included in the Effectiveness Population. This retreated/redosed treatment group comprised 87 participants that received their second treatment course of EN3835 in Study EN3835-202 having received their first treatment course in Study EN3835-201 and 75 participants that received both their first and second treatment courses in Study EN3835-202. Treatment phase is defined as the time period from the second EN3835 treatment date to the End of Study EN3835-202.
Time Frame: Day 71 - Day 360
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 162
Participants
  Second EN3835 Treatment: Treatment Day 71: number analyzed (Participants) | 159
  Second EN3835 Treatment: Treatment Day 71: Very Much Improved (3) | 16
  Second EN3835 Treatment: Treatment Day 71: Much Improved (2) | 33
  Second EN3835 Treatment: Treatment Day 71: Improved (1) | 69
  Second EN3835 Treatment: Treatment Day 71: No Change (0) | 32
  Second EN3835 Treatment: Treatment Day 71: Worse (-1) | 7
  Second EN3835 Treatment: Treatment Day 71: Much Worse (-2) | 1
  Second EN3835 Treatment: Treatment Day 71: Very Much Worse (-3) | 1
  Second EN3835 Tx: Treatment Observation Day 360: number analyzed (Participants) | 143
  Second EN3835 Tx: Treatment Observation Day 360: Very Much Improved (3) | 16
  Second EN3835 Tx: Treatment Observation Day 360: Much Improved (2) | 14
  Second EN3835 Tx: Treatment Observation Day 360: Improved (1) | 64
  Second EN3835 Tx: Treatment Observation Day 360: No Change (0) | 39
  Second EN3835 Tx: Treatment Observation Day 360: Worse (-1) | 7
  Second EN3835 Tx: Treatment Observation Day 360: Much Worse (-2) | 3
  Second EN3835 Tx: Treatment Observation Day 360: Very Much Worse (-3) | 0

15. Secondary Outcome: Subject Satisfaction With EFP Treatment at the End of Study (EOS) in Observation Phase, Observation Visit Day 360
Description: Subject Satisfaction with Cellulite Treatment Scale is a 5-level scale designed for participants to assess their satisfaction with cellulite treatment. The scale ranges from "+2" (I am very satisfied with the cellulite treatment on my buttocks or thighs) to "-2" (I am very dissatisfied with the cellulite treatment on my buttocks or thighs). Percentages are based on the number of evaluable participants at each visit. Observation Phase is defined as the time period from Screening to the first treatment date of the same treatment area in Study EN3835-202, or the end of Study EN3835-202 if there was no treatment received for the same treatment area in Study EN3835-202. (EFP = Edematous Fibrosclerotic Panniculopathy, aka Cellulite)
Time Frame: Day 360
Population: Observation Population included all participants who rolled over from Study EN3835-201
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 97 | 19
Participants
  Very Satisfied with Treatment (2) | 14 | 0
  Satisfied with Treatment (1) | 41 | 4
  Neither Dissatisfied nor Satisfied with Tretmt (0) | 23 | 11
  Dissatisfied with Treatment (-1) | 14 | 4
  Very Dissatisfied with Treatment (-2) | 5 | 0

16. Secondary Outcome: Subject Satisfaction With EFP Treatment in Treatment Phase for Subjects With Second EN3835 Treatment
Description: Subject Satisfaction with Cellulite Treatment Scale is a 5-level scale designed for participants to assess their satisfaction with cellulite treatment. The scale ranges from "+2" (I am very satisfied with the cellulite treatment on my buttocks or thighs) to "-2" (I am very dissatisfied with the cellulite treatment on my buttocks or thighs). Percentages are based on the number of evaluable participants at each visit. One hundred sixty-two participants received a second treatment course in Study EN3835-202 and were included in the Effectiveness Population. This retreated/redosed treatment group comprised 87 participants that received their second treatment course of EN3835 in Study EN3835-202 having received their first treatment course in Study EN3835-201 and 75 participants that received both their first and second treatment courses in Study EN3835-202. Treatment phase is defined as the time period from the second EN3835 treatment date to the End of Study EN3835-202.
Time Frame: Day 71 - Day 360
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 162
Participants
  Second EN3835 Treatment: Treatment Day 71: number analyzed (Participants) | 159
  Second EN3835 Treatment: Treatment Day 71: Very Satisfied wth Treatment (2) | 34
  Second EN3835 Treatment: Treatment Day 71: Satisfied with Treatment (1) | 67
  Second EN3835 Treatment: Treatment Day 71: Neither Dissatisfied nor Satisfied with Tx (0) | 36
  Second EN3835 Treatment: Treatment Day 71: Dissatisfied with Treatment (-1) | 13
  Second EN3835 Treatment: Treatment Day 71: Very Dissatisfied with Treatment (-2) | 9
  Second EN3835 Treatment: Treatment Obsv Day 360: number analyzed (Participants) | 143
  Second EN3835 Treatment: Treatment Obsv Day 360: Very Satisfied wth Treatment (2) | 25
  Second EN3835 Treatment: Treatment Obsv Day 360: Satisfied with Treatment (1) | 50
  Second EN3835 Treatment: Treatment Obsv Day 360: Neither Dissatisfied nor Satisfied with Tx (0) | 45
  Second EN3835 Treatment: Treatment Obsv Day 360: Dissatisfied with Treatment (-1) | 16
  Second EN3835 Treatment: Treatment Obsv Day 360: Very Dissatisfied with Treatment (-2) | 7

17. Other Pre Specified Outcome: Overall Serum Antibody at Observation Visit Day 360
Description: Percent of participants that are seropositive. Descriptive statistics are based on log10 transformation of titer levels. Percent is based on the number of subjects who had immunogenicity lab samples drawn at the visit
Time Frame: Day 360
Population: Observation Population included all participants who rolled over from Study EN3835-201 (259 participants in Observation Phase). Included all participants with collected samples at Day 360.
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 19 | 4
Participants
  anti-AUX-I: Observation Visit Day 360: Seropositive | 17 | 2
  anti-AUX-I: Observation Visit Day 360: Seronegative | 2 | 2
  anti-AUX-II: Observation Visit Day 360: Seropositive | 16 | 2
  anti-AUX-II: Observation Visit Day 360: Seronegative | 3 | 2

18. Other Pre Specified Outcome: Overall Antibody Log Titer Levels at Observation Visit Day 360
Description: Descriptive statistics are based on log10 transformation of titer levels.
Time Frame: Day 360
Population: Observation Population included all participants who rolled over from Study EN3835-201 (all 259 participants that rolled over in Observation Phase). Included Seropositive participants at Day 360.
Measure: Mean (Standard Deviation); unit: log 10 titer
Arm/Group | EN3835 0.84 mg | Placebo
Number analyzed (Participants) | 17 | 2
log 10 titer
  anti-AUX-I: Observation Visit Day 360 positive | 3.085 (1.192) | 2.576 (0.213)
  anti-AUX-II: Observation Visit Day 360 positive: number analyzed (Participants) | 16 | 2
  anti-AUX-II: Observation Visit Day 360 positive | 3.175 (1.239) | 1.547 (0.315)

19. Other Pre Specified Outcome: Neutralizing Antibodies at Observation Visit Day 360
Description: Participants with binding antibodies were tested for neutralizing antibodies.
Time Frame: Day 360
Population: Observation Population included all participants who rolled over from Study EN3835-201 (259 participants in Observation Phase).Included Seropositive participants at Day 360.
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 23
Participants
  Neutralizing AUX-I Antibody: number analyzed (Participants) | 18
  Neutralizing AUX-I Antibody: Negative | 5
  Neutralizing AUX-I Antibody: Positive | 13
  Neutralizing AUX-II Antibody: Negative | 14
  Neutralizing AUX-II Antibody: Positive | 9

20. Other Pre Specified Outcome: Overall Antibody Log Titer Levels by Visit During the Treatment Phase for Participants With a Second EN3835 Treatment
Description: Descriptive statistics are based on Seropositive participants. Descriptive statistics are based on log10 transformation of titer levels.
Time Frame: Day 1 to Day 360
Population: Safety Population included participants with seropositive antibody results
Measure: Mean (Standard Deviation); unit: Log 10 titer
Groups:
- EN3835 Treatment Regions: Buttocks & Thighs Treatment Regions Treated with EN3835 0.84mg Collagenase Clostridium Histolyticum
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 163
Log 10 titer
  anti-AUX-I: Treatment Day 1 positive: number analyzed (Participants) | 152
  anti-AUX-I: Treatment Day 1 positive | 4.038 (0.697)
  anti-AUX-I: Treatment Day 71 positive: number analyzed (Participants) | 151
  anti-AUX-I: Treatment Day 71 positive | 6.268 (0.786)
  anti-AUX-I: Treatment Observation Day 360 positive: number analyzed (Participants) | 139
  anti-AUX-I: Treatment Observation Day 360 positive | 4.964 (0.584)
  anti-AUX-II: Treatment Day 1 positive: number analyzed (Participants) | 152
  anti-AUX-II: Treatment Day 1 positive | 3.853 (0.854)
  anti-AUX-II: Treatment Day 71 positive: number analyzed (Participants) | 151
  anti-AUX-II: Treatment Day 71 positive | 5.832 (0.736)
  anti-AUX-II: Treatment Observation Day 360 positiv: number analyzed (Participants) | 139
  anti-AUX-II: Treatment Observation Day 360 positiv | 4.714 (0.635)

21. Other Pre Specified Outcome: Neutralizing Antibodies in Treatment Phase for Participants With a Second EN3835 Treatment
Description: Tx Obs = Treatment Observation
Time Frame: Day 71 to Day 360
Population: Safety Population included participants with observed antibody levels at Day 71 in Q1 and Q4
Measure: Count of Participants; unit: Participants
Arm/Group | EN3835 Treatment Regions
Number analyzed (Participants) | 38
Participants
  Treatment Day 71: Neutralizing AUX-I Antibody: Negative | 2
  Treatment Day 71: Neutralizing AUX-I Antibody: Positive | 36
  Treatment Day 71: Neutralizing AUX-II Antibody: number analyzed (Participants) | 35
  Treatment Day 71: Neutralizing AUX-II Antibody: Negative | 10
  Treatment Day 71: Neutralizing AUX-II Antibody: Positive | 25
  Tx Obs Day 360: Neutralizing AUX-I Antibody: number analyzed (Participants) | 36
  Tx Obs Day 360: Neutralizing AUX-I Antibody: Negative | 21
  Tx Obs Day 360: Neutralizing AUX-I Antibody: Positive | 15
  Tx Obs Day 360: Neutralizing AUX-II Antibody: number analyzed (Participants) | 35
  Tx Obs Day 360: Neutralizing AUX-II Antibody: Negative | 32
  Tx Obs Day 360: Neutralizing AUX-II Antibody: Positive | 3

ADVERSE EVENTS:
Time Frame: All (serious or nonserious) AEs, from Day 1 up to Day 720 (720 days after first exposure to study drug in predecessor study EN3835-201)
Description: All (serious and nonserious) AEs, whether elicited or observed during study visits or spontaneously reported by the participant, including events that occurred from the time the participant signed the study-specific consent form until completion of or discharge from the study.
  One death due to a motor vehicle accident reported in the Treatment Phase in a subject treated with EN3835 that was assessed as not related to EN3835.
Groups:
- Observation Phase: Observation of Buttock or Thigh Treated with EN3835: 0.84mg Collagenase Clostridium Histolyticum or with Placebo in Study EN3835-201
- EN3835 Treatment Phase: Buttock or Thigh Treated with EN3835: 0.84mg Collagenase Clostridium Histolyticum
Arm/Group | Observation Phase | EN3835 Treatment Phase
All-Cause Mortality (participants affected / at risk) | 0/259 | 1/200
Serious Adverse Events (participants affected / at risk) | 1/259 | 4/200
Other Adverse Events (participants affected / at risk) | 0/259 | 176/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Observation Phase (N=259) | EN3835 Treatment Phase (N=200)
Appendicitis (Infections and infestations) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spontaneous Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Hypertensive Urgency (Vascular disorders) | 0 | 1
Death from Motor Vehicle Accident (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Observation Phase (N=259) | EN3835 Treatment Phase (N=200)
Injection site bruising (General disorders) | 0 | 170
Injection site pain (General disorders) | 0 | 113
Injection site nodule (General disorders) | 0 | 39
Injection site pruritus (General disorders) | 0 | 33
Injection site swelling (General disorders) | 0 | 19
Injection site discolouration (General disorders) | 0 | 18
Upper respiratory tract infection (Infections and infestations) | 0 | 11 — No AEs occurred at a frequency greater than or equal to 5% in Observation Phase

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/60/NCT02942160/Prot_SAP_000.pdf